CLINICAL TRIAL: NCT04438876
Title: The Effects of Functional Power Training on Frail and Pre-frail Community - Dwelling Older Adults in Singapore: A Randomised Controlled Trial
Brief Title: The Effects of Functional Power Training on Frail and Pre-frail Community - Dwelling Older Adults in Singapore
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geriatric Education and Research Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: GERI1618
Record Dates: First submitted 2020-06-15; First posted 2020-06-19 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2020-06

CONDITIONS: Frailty; Muscle Weakness
MeSH Terms: conditions — Frailty; Muscle Weakness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Function power training (Experimental): 12-week structured FPT program, conducted by a certified trainer from a community service provider. Sessions were held twice weekly at the respective community senior activity centers, each lasting 60 minutes in duration.
  Interventions: Other: Functional Power Training
- Usual care (Active Comparator): Participants either continued the usual exercise program provided by their respective community senior activity centers or their personal exercise routine.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Functional Power Training — The exercise intervention encompassed high-velocity movement, balance, and mobility exercises with the use of body weight and resistance bands as resistance. Participants were instructed to move rapidly during the concentric phase and slowly during the eccentric phase when performing the dynamic exercises.
  Arms: Function power training
Other: Usual care — Participants either continued the usual exercise program provided by their respective community senior activity centers or their personal exercise routine.
  Arms: Usual care

SUMMARY:
To investigate the efficacy of a 12-week Functional Power Training (FPT) program in pre-frail and frail community-dwelling older adults in Singapore for the management of physical frailty. The proposed study will provide information on the benefits of FPT on physical performances of older adults and help to shape future exercise recommendations to slow or reverse the onset and severity of physical frailty.

ELIGIBILITY:
Inclusion Criteria:

* aged 55 years and above
* low muscle strength - handgrip strength less than 26kg for men and 18kg for women
* ambulate without human assistance
* able to understand basic instructions

Exclusion Criteria:

* currently enrolled in another study
* acute musculoskeletal injury
* unable to participate in the full duration of the study
* unwilling to participate if not assigned to the intervention group
* deemed not suitable to participate in exercise by a medical doctor

Ages: 55 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change of Frail status at 12 and 24 weeks | baseline, 12 weeks, 24 weeks
  Cardiovascular Health Study (CHS) Frailty status which characterizes frailty based on five components: unintentional weight loss, weakness, slowness, exhaustion and low physical activity. 1 point for each category. Robust: 0 point, Pre-Frail: 1-2 points , Frail: 3-5 points.
Change of hand grip strength at 12 and 24 weeks | baseline, 12 weeks, 24 weeks
  Hand grip strength (kg)
Change of knee extensor strength at 12 and 24 weeks | baseline, 12 weeks, 24 weeks
  Knee extensor strength (kg)
Change of Timed up and go (TUG) at 12 and 24 weeks | baseline, 12 weeks, 24 weeks
  Timed up and go (TUG) (seconds)
Change of SPPB at 12 and 24 weeks | baseline, 12 weeks, 24 weeks
  Short Physical Performance Battery (SPPB) consist of:
  1. Balance test
  2. Gait speed
  3. Chair stand test

SECONDARY OUTCOMES:
Exercise adherence | baseline, 12 weeks, 24 weeks
  Exercise journals

CONTACTS AND LOCATIONS:
Overall Officials: Shiou-Liang Wee, PhD, Principal Investigator — Geriatric Education & Research Institute
Locations (1):
- Geriatric Education & Research Institute, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tou NX, Wee SL, Seah WT, Ng DHM, Pang BWJ, Lau LK, Ng TP. Effectiveness of Community-Delivered Functional Power Training Program for Frail and Pre-frail Community-Dwelling Older Adults: a Randomized Controlled Study. Prev Sci. 2021 Nov;22(8):1048-1059. doi: 10.1007/s11121-021-01221-y. Epub 2021 Mar 19. PMID 33742266